CLINICAL TRIAL: NCT04653246
Title: Phase 2, Multi-Center, Single-Arm, Open-Label Study to Evaluate the Efficacy and Safety of the Combination Regimen Isatuximab, Lenalidomide, Bortezomib, and Dexamethasone in Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Isatuximab, Lenalidomide, Bortezomib, and Dexamethasone in NDMM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jacob Laubach, MD (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Jacob Laubach, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-207
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma; Newly Diagnosed Multiple Myeloma (NDMM); Autologous Stem Cell Transplant
Keywords: Multiple Myeloma; Newly diagnosed multiple myeloma (NDMM); Autologous stem cell transplant (ASCT).; High dose therapy (HDT)
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab; Lenalidomide; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Isa-RVD (Experimental): The main study consists of 4 phases a) 28-day screening phase; b) an induction phase inclusive of two 42-day induction treatment cycles: Isatuximab (IV), Bortezomib (SQ). Lenalidomide (PO), Dexamethasone; c) Followed by stem cell mobilization (at the discretion of the Principal Investigator [PI]);d) Participants will proceed with either autologous stem cell transplant or two additional induction cycles.
  - Induction will be followed by a maintenance phase that continues until disease progression.
  Interventions: Drug: Isatuximab; Drug: Lenalidomide; Drug: Bortezomib Injection; Drug: Dexamethasone

INTERVENTIONS:
Drug: Isatuximab — Via IV at predetermined dosage and predetermined days during each cycle
  Other Names: Sarclisa
Drug: Lenalidomide — Oral, predetermined dosage and predetermined days during each cycle
  Other Names: Revlimid
Drug: Bortezomib Injection — SQ Oral, predetermined dosage and predetermined days during each cycle
Drug: Dexamethasone — IV or Oral predetermined dosage and predetermined days during each cycle

SUMMARY:
This research is testing whether the investigational drug isatuximab is safe and effective when used in combination with standard agents for the treatment of newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
This is a multi-center, single-arm, open-label, Phase 2 study in patients with newly diagnosed multiple myeloma (NDMM) eligible for high dose therapy (HDT) and autologous stem cell transplant (ASCT).

In this research study, investigators are evaluating whether isatuximab is safe and effective in participants with newly diagnosed multiple myeloma when given in combination with lenalidomide, bortezomib, and dexamethsone.

* This research study involves administration of a four-drug chemotherapy regimen that combines the Investigational drug isatuximab with a standard chemotherapy regimen comprised of lenalidomide, bortezomib, and dexamethasone.
* This 4-drug regimen is not considered standard of the treatment of newly diagnosed multiple myeloma.

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug or combination of drugs to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The U.S. Food and Drug Administration (FDA) has approved lenalidomide, bortezomib, and dexamethasone as treatment options for this disease but the combination of these agents with isatuximab hasn't been approved.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed with MM based on standard IMWG criteria and currently requires treatment.
* Provided voluntary written informed consent before performance of any study-related procedures not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care
* Age ≤ 75 years, with patients over the age of 70 requiring PI approval
* Measurable disease defined as at least one of the following:

  * Serum M protein ≥ 0.5 g/dL (≥5 g/L)
  * Urine M protein ≥ 200 mg/24 hours
  * Serum free light chain (FLC) assay: Involved FLC assay ≥10 mg/dL (≥100 mg/L) and an abnormal serum FLC ratio (<0.26 or >1.65)
* Screening Laboratory evaluations within the following parameters

  * Absolute neutrophil count (ANC) ≥ 1,000 cells/dL (1.0 x 109/L) (Growth factors cannot be used within 14 days before first drug administration)
  * Platelet count ≥ 75,000 cells/dL (75 x 109/L) if < 50% BM nucleated cells are plasma cells, ≥ 30,000 cells/dL if ≥ 50% of BM nucleated cells are plasma cells. (without transfusions required during the 3 days prior to the screening hematologic test)
  * Total Bilirubin ≤ 2.0 X upper limit of normal (ULN) (except patients with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
  * AST (SGOT) and ALT (SGPT) ≤ 3.0 x ULN
  * Calculated creatinine clearance ≥ 30 mL/min
  * Hemoglobin ≤ 8 g/dL
* ECOG performance status ≤ 2 (Appendix A)
* Participant agrees to be registered into the mandatory Revassist REMS® program, and be willing and able to comply with the requirements of the RevAssist REMS® program.
* Ability to understand and the willingness to sign a written informed consent document
* Participant is considered eligible for ASCT by the treating physician.

Exclusion Criteria:

* Prior therapy for multiple myeloma
* Diagnosed or treated for another malignancy within 3 years prior to enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in-situ malignancy, or low risk prostate cancer after curative therapy.
* Central nervous system involvement.
* Peripheral neuropathy ≥ Grade 3, or Grade 2 with pain on clinical examination during the screening period.
* Any medical or psychiatric illness that in the Investigator's opinion, would impose excessive risk to the patient or would adversely affect his/her participating in this study.
* Concurrent uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, Grade 3 thromboembolic event or myocardial infarction within the past 6 months.
* Prior major surgical procedure or radiation therapy within 4 weeks of initiation of therapy (this does not include limited course of radiation used for management of bone pain within 7 days of initiation of therapy).
* Daily requirement for corticosteroids (equivalent to > 10 mg/day prednisone for more than 7 days (except for inhalation corticosteroids).
* Concurrent symptomatic amyloidosis or plasma cell leukemia
* POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin changes)
* Known active infection requiring parenteral or oral anti-infective treatment within 14 days of start of therapy.
* Active hepatitis B or hepatitis C viral infection
* Pregnant or breastfeeding female or female who intends to become pregnant during the participation in the study. Females of childbearing potential (FCBP) unwilling to prevent pregnancy by the use of 2 reliable methods of contraception for ≥4 weeks before the start of study treatment, during treatment (including dose interruptions), and up to 3 months following the last dose of study treatment and/or who are unwilling or unable to be tested for pregnancy before study treatment initiation (2 negative tests), weekly during 1st month of treatment and then prior each treatment cycle administration or every 2 weeks in case or irregular menstrual cycles up to 3 months following the last dose of study treatment.
* Male participants who disagree to practice true abstinence or disagree to use a condom during sexual contact with a pregnant female or a FCBP while participating in the study, during dose interruptions and at least 3 months following study treatment discontinuation, even if has undergone a successful vasectomy.

  * Note 1: a FCBP is a female who: 1) has achieved menarche at some time point, 2) has not undergone a hysterectomy or bilateral oophorectomy or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months).
  * Note 2: True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Receiving any other investigational agents
* Inability to tolerate thromboprophylaxis
* Hypersensitivity (or contraindication) to dexamethasone, sucrose histidine (as base and hydrochloride salt), boron, mannitol, and polysorbate 80, or to any of the components of the study therapy
* Hypersensitivity to steroids or H2 blockers that would prohibit further treatment with these agents.

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2029-01-13 (Estimated)

PRIMARY OUTCOMES:
stringent Complete Response (sCR) | 84 days
  proportion of patients who have achieved sCR, according to IMWG criteria, by the end of two cycles of induction treatment. Response will be evaluated using a Simon optimal two-stage design.

SECONDARY OUTCOMES:
Time to Progression | time from registration to progression, censored at date last known to be progression-free for those who have not progressed and censored at time of death up to 42 months
  Progression-free probabilities over time will be estimated using the Kaplan-Meier method (Kaplan, 1958), presenting an estimate of median time to progression (TTP) with 95% confidence intervals (CIs). Time to progression is defined as time from registration to progression, censored at date last known to be progression-free for those who have not progressed and censored at time of death for those who died.
Progression Free Survival | time from registration to disease progression or death from any cause, censored at date last known to be progression-free for those who have not progressed or died up to 42 months
  - Progression-free survival (PFS) will be analyzed similarly to time to progression: Progression-free probabilities over time will be estimated using the Kaplan-Meier method (Kaplan, 1958), presenting an estimate of median Time to progression (TTP) with 95% confidence intervals (CIs Time from registration to disease progression or death from any cause, censored at date last known to be progression-free for those who have not progressed or died
Duration of Response | Time from first response after treatment to the date of disease progression or death from any cause, or date last known progression-free and alive for those who have not progressed or died up to 42 months
  Duration of Response will be analyzed similarly to time to progression: Progression-free probabilities over time will be estimated using the Kaplan-Meier method (Kaplan, 1958), presenting an estimate of median time to progression (TTP) with 95% confidence intervals (CIs Time from first response after treatment to the date of disease progression or death from any cause, or date last known progression-free and alive for those who have not progressed or died.
Overall Survival | Overall survival: time from registration to death from any cause or date last known alive for those who have not died up to 42 months
  Overall Survival will be analyzed similarly to time to progression: Progression-free probabilities over time will be estimated using the Kaplan-Meier method (Kaplan, 1958), presenting an estimate of median time to progression (TTP) with 95% confidence intervals (CIs
  Overall survival: time from registration to death from any cause or date last known alive for those who have not died
Number of Participants with Treatment Related Adverse Events as Assessed by CTCAE v 5.0 | Induction to up to 3.5 years
  Common Terminology Criteria for Adverse Events (CTCAE) of the National Cancer Institute (NCI) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jacob C Laubach, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu